CLINICAL TRIAL: NCT03396718
Title: De-escalation of Adjuvant Radio (Chemo) Therapy for HPV-positive Head and Neck Squamous Cell Carcinomas: A Phase I Study to Reduce Late Toxicity
Brief Title: De-escalation of Adjuvant Radio (Chemo) Therapy for HPV-positive Head-neck Squamous Cell Carcinomas
Acronym: DELPHI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other); National Center for Tumor Diseases (NCT) Dresden (Unknown); National Center for Tumor Diseases, Heidelberg (Other); Radiation Oncology Working Group of the German Cancer Society (Other)
Responsible Party: Principal Investigator, Mechthild Krause, Director of the Department of Radiotherapy and Radiation Oncology, Technische Universität Dresden
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STR-DELPHI-2016
Record Dates: First submitted 2017-10-24; First posted 2018-01-11 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Head-and-neck Squamous Cell Carcinoma
Keywords: Head and neck cancer; Oropharyngeal cancer; postoperative; radiotherapy; radiochemotherapy; de-intensification; HPV
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms; Oropharyngeal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Interventional Arm A - HPV(+) (Experimental): De-escalation Radio(chemo)therapy - Level 1
  Interventions: Radiation: De-escalation radio(chemo)therapy - Level 1
- Interventional Arm B - HPV(+) (Experimental): De-escalation Radio(chemo)therapy - Level 2
  Interventions: Radiation: De-escalation radio(chemo)therapy - Level 2
- Observational Arm A - HPV(-) (Active Comparator): Standard Radio(chemo)therapy
  Interventions: Radiation: Standard radio(chemotherapy)
- Observational Arm B - HPV(+) (Active Comparator): Standard Radio(chemo)therapy
  Interventions: Radiation: Standard radio(chemotherapy)

INTERVENTIONS:
Radiation: De-escalation radio(chemo)therapy - Level 1 — 55/ 59,4 Gy (intermediate / high risk group)
  Arms: Interventional Arm A - HPV(+)
Radiation: De-escalation radio(chemo)therapy - Level 2 — 48,4/ 55 Gy (intermediate / high risk group)
  Arms: Interventional Arm B - HPV(+)
Radiation: Standard radio(chemotherapy) — 60/ 66 Gy (intermediate / high risk group)
  Arms: Observational Arm A - HPV(-); Observational Arm B - HPV(+)

SUMMARY:
In patients with squamous cell carcinoma of the oral cavity, the oropharynx and larynx with local advanced tumors (pathologic stage T3 = pT3) and or lymph node involvement (pN+) postoperative radio - or radiochemotherapy is the standard of care. Postoperative radiochemotherapy is indicated in patients with multiple lymph node metastasis, lymph node metastasis with extracapsular spread and / or residual tumor (R1-Status) after resection. Oropharyngeal cancer caused by HPV (human papillomavirus 16) is a distinct subgroup with a known sensitivity to radiotherapy (RTx) or radiochemotherapy (RCTx). Additionally a superior outcome after R(C)Tx over HPV negative patients was shown for patients treated with primary or adjuvant RCTx. To date it is unknown if the total dose of the radiotherapy can be safely reduced with the aim to decrease the therapy associated late effects.

Patients with a HPV associated carcinoma that take part in the study will be treated with a reduced radiotherapy dose, chemotherapy will be prescribed based on clinical factors (number of affected lymph node, presence of extracapsular spread or residual tumor). Radiation dose will be reduced in two steps.

DETAILED DESCRIPTION:
For all patients taking part in the study the HPV status of the resected tumor will be determined centrally by p16 immunohistochemistry and confirmation will be done by HPV DNA assessment using Polymerase Chain Reaction (PCR)-based array. Patients positive for HPV will be treated with a reduced RT dose to the tumor and to elective neck. HPV negative patients will be treated with standard radio- or radiochemotherapy. Patients deemed at high risk for locoregional recurrences (presence of extracapsular spread, residual tumor or multiple affected nodes) will be treated separately from patients deemed at intermediate risk (T>=3, and / or 1-3 nodes positive). The high risk group will be treated with a higher dose and concurrent chemotherapy. After inclusion of 30 patients per treatment group, follow up for the first 10 patients of the of the first de-escalation level will be awaited for two years and safety of the intervention will be assessed. The second de-escalation level will only be opened for accrual if less than 2 locoregional recurrences will occur within the first 10 patients per treatment group.

ELIGIBILITY:
Inclusion Criteria:

* Condition after surgical removal of a squamous cell carcinoma of the oropharynx and adequate lymph node dissection
* Indication for adjuvant radiotherapy or radiochemotherapy in the interdisciplinary tumor board
* Good general state (ECOG performance status 0 or 1)
* Adequate compliance to ensure closely follow-up
* Patient's consent and written consent
* Neck dissection of at least the tumor bearing side

Additional Inclusion Criteria Arm intermediate risk (at least one of the criteria must be fulfilled):

* pT3 and R0 and / or
* histologically confirmed involvement of lymph nodes (n = 1-3) and no extracapsular extension of the lymph node metastasis

Additional Inclusion Criteria Arm high risk (at least one of the criteria must be fulfilled):

* residual tumor (R1 status) and / or
* pathologic stage T4 (pT4) status and / or
* more than 3 infected lymph nodes and / or
* extracapsular extension of at least one lymph node metastasis

Exclusion Criteria:

* Patients with a cumulative nicotine abuse > 30 packyears. These patients are not included in the intervention arms, but are always included in the observation arms (regardless of HPV status).
* radiologically presumed or histologically confirmed distant metastasis
* R2 resection or macroscopically visible residual tumor after surgery
* no neck dissection
* interval between last operation and planned irradiation start > 7 weeks
* contraindication against a guideline-appropriate adjuvant radiation or radiochemotherapy according to the clinical risk constellation
* tumor disease in the last five years before the beginning of the study (except basaliomas of the skin, in-situ carcinoma of the cervix uteri or breast, or tumors with similar prognosis which are considered to be very likely to be cured)
* malignant tumor disease in the head and neck region, regardless of interval and prognosis
* Pre-irradiation with risk of dose overlap
* participation in another clinical trial if further experimental therapy is necessary or the treatments/ protocols are mutually exclusive (e.g. altered chemotherapy, additional consolidation chemotherapy). Allowed is the additional participation in observation studies or supportive therapy studies.
* diseases or conditions which do not allow the person concerned to assess the nature and scope and possible consequences of the clinical trial
* pregnant or lactating women
* evidence that the participant is not expected to comply with the study protocol (e.g. lack of cooperation)
* missing written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2018-11-29 (Actual); Primary Completion 2029-11-30 (Estimated); Study Completion 2032-11-30 (Estimated)

PRIMARY OUTCOMES:
rate of locoregional recurrences | 24 months after end of treatment
  measured from the last day of treatment

SECONDARY OUTCOMES:
overall survival | 60 months and 5 years after end of treatment
  measured from the last day of treatment
acute toxicity | 3 months after end of treatment
  The occurrence of acute side effects (up to 90 days after start of treatment) will be recorded and documented based on CTCAE 4.0.
late toxicity | 24 months after end of treatment
  The occurrence of late side effects will be recorded and documented based on CTCAE 4.0 after every follow-up visit.
quality of life of cancer patients | 24 months after end of treatment
  The assessment of quality of life (QoL) is carried out using the EORTC quality of life questionnaire (QLQ) C30. Quality of life will be documented immediately before the start of therapy, after completion of postoperative radiotherapy and at every follow-up visit. QOL will be measured as change from baseline over time.
quality of life - disease specific | 24 months after end of treatment
  The assessment of quality of life (QOL) is carried out using the EORTC quality of life questionnaire (QLQ) disease-specific module for head and neck cancer H&N35. Quality of life will be documented immediately before the start of therapy, after completion of postoperative radiotherapy and at every follow-up visit. QOL will be measured as change from baseline over time.
rate of locoregional recurrences | 5 years after end of treatment
  measured from the last day of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Mechthild Krause, Prof., Study Chair — University of Technology, University Hospital Carl Gustav Carus, Department of Radiation Therapy and Radiation Oncology, German Consortium for Translational Cancer Research (DKTK)
Locations (10):
- Germany (10):
  - University Clinic Tübingen, Tübingen, Baden-Wurttemberg
  - University Clinic Essen, Essen, North Rhine-Westphalia
  - University Clinic Dresden, Dresden, Saxony
  - Charité - Universitätsmedizin Berlin, Berlin
  - University Clinic Frankfurt, Frankfurt am Main
  - University Clinic Freiburg, Freiburg im Breisgau
  - University Clinic Heidelberg, Heidelberg
  - LMU Munich University Hospital, München
  - TUM University Hospital, München
  - University Clinic Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: No